CLINICAL TRIAL: NCT01431183
Title: Seasonal Influenza Vaccination Reminders for Children With High-risk Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Kevin Dombkowski, Research Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 5U01IP000132 (NIH)
Record Dates: First submitted 2011-09-06; First posted 2011-09-09 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Seasonal Influenza Vaccination
Keywords: influenza; vaccine; reminder / recall; immunization registry; immunization information systems
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- mailed reminder notice (Active Comparator): Seasonal influenza vaccination reminder sent by postal mail
  Interventions: Behavioral: Mailed influenza vaccination reminder notice
- No reminder notice (No Intervention): No seasonal influenza vaccination reminder sent by postal mail

INTERVENTIONS:
Behavioral: Mailed influenza vaccination reminder notice — Influenza vaccination reminder sent by postal mail
  Arms: mailed reminder notice

SUMMARY:
The objective of this study was to assess the feasibility and effectiveness of using a statewide immunization information system (IIS) to send seasonal influenza vaccine reminders from Local Health Departments (LHDs), targeting children with high-risk conditions.

ELIGIBILITY:
Inclusion Criteria:

* children, 24-60 months
* current or previous enrollment in Medicaid (Michigan)
* presence of at least 1 chronic condition, as indicated by the Michigan Care Improvement Registry (MCIR)
* resident of Kalamazoo, Ottawa, or Kent counties (Michigan)

Exclusion Criteria:

* receipt of influenza prior to notification date
* ineligible for reminder/recall notification in the Michigan Care Improvement Registry (MCIR)

Ages: 24 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3618 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
seasonal influenza vaccination | up to 4 months following reminder notification
  Receipt of 1 or more dose of seasonal influenza vaccine, either trivalent inactivated influenza vaccine (TIV) or live attenuated influenza vaccine (LAIV)

SECONDARY OUTCOMES:
invalid mailing address | up to 4 months following reminder notification
  Postal mailing address determined to be invalid for mail delivery, either by physical return of mailed reminder notification, or through the United States Postal Service's National Change of Address (NCOA) process

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Dombkowski, DrPH, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Child Health Evaluation and Research Unit, Ann Arbor, Michigan, United States

REFERENCES:
- [Derived] Dombkowski KJ, Harrington LB, Dong S, Clark SJ. Seasonal influenza vaccination reminders for children with high-risk conditions: a registry-based randomized trial. Am J Prev Med. 2012 Jan;42(1):71-5. doi: 10.1016/j.amepre.2011.09.028. PMID 22176850